CLINICAL TRIAL: NCT05791396
Title: Efficacy and Mechanisms of Fecal Microbiota Transplantation to Eradicate Intestinal Colonization by Carbapenem-resistant Enterobacteriaceae
Brief Title: FMT to Eradicate Intestinal Colonization by Carbapenem-resistant Enterobacteriaceae
Acronym: FMT_CRE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Cammarota Giovanni, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5544
Record Dates: First submitted 2023-03-16; First posted 2023-03-30 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Enterobacteriaceae Infections; Multi-antibiotic Resistance
Keywords: Fecal microbiota transplantation; Enterobacteriaceae; Multi-drug resistant bacteria
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To mask treatments to physicisans and recipients, both FMT bottles and syringes will be covered with dark-coloured paper before the infusion, and the patients will be unable to see the endoscopic display during the procedure. Moreover, the physicians who will evaluate patients at follow-up will not aware of the treatment being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor FMT (Experimental): Patients enrolled in this arm will receive donor FMT
  Interventions: Biological: Donor - FMT
- Placebo FMT (Placebo Comparator): Patients enrolled in this arm will receive placebo FMT (that will be made of water)
  Interventions: Other: Placebo FMT

INTERVENTIONS:
Biological: Donor - FMT — this intervention is represented by the administration, in the recipients' gut, of donor microbiota through FMT
  Arms: Donor FMT
Other: Placebo FMT — This intervention is represented by the administration, in the recipients' gut, of a placebo through colonoscopy
  Arms: Placebo FMT

SUMMARY:
Antibiotic resistance (AR) is a critical public health threat and one of the greatest challenges of the 21st century. In an estimate of 2019, nearly 700.000 infections and 33.000 attributable deaths from multi-drug-resistant bacteria (MDRB) have occurred in Europe in 2015. The gastrointestinal tract is a large reservoir for MDRB, and the gut microbiota can harbor a collection of AR genes, called gut resistome. Preliminary nonrandomized evidence suggests that fecal microbiota transplant (FMT) could be a promising treatment option to eradicate MDRB, but established evidence, as well as mechanisms that underpin this therapeutic pathway, are still unavailable. Leveraging our expertise in FMT (OU1), microbiome (OU2) and MDRB (OU3), we aim to evaluate the efficacy of FMT (from donors with limited presence of AR genes) in eradicating intestinal MDRB through a randomized controlled trial and identifying microbial features that are associated with clinical efficacy and clearance of AR genes

DETAILED DESCRIPTION:
Antibiotic resistance (AR) is a critical public health threat and one of the greatest challenges of the 21st century. In an estimate of 2019, nearly 700.000 infections and 33.000 attributable deaths from multi-drug-resistant bacteria (MDRB) have occurred in Europe in 2015. Despite specific interventions, including antibiotic stewardship measures and AR surveillance programs, this burden has nearly doubled since 2007 and is highest for infections caused by intestinal bacteria. The gastrointestinal tract is a large reservoir for MDRB, and the gut microbiota can harbor a collection of AR genes, called gut resistome. There is increasing evidence that healthy gut microbiota can prevent the colonization of MDRB through mechanisms of colonization resistance, including competition, production of antimicrobial peptides, immune regulation. However, this protective mechanism can be impaired by therapies that alter gut microbiota (e.g. antibiotics). The restoration of healthy gut microbiota by fecal microbiota transplantation (FMT) may lead to the eradication of antibiotic-resistant bacteria. After becoming a standard treatment for Clostridioides difficile infection, FMT has been investigated in several disorders, and preliminary nonrandomized reports suggest that it could be a promising treatment option to eradicate MDRB, but established evidence, as well as mechanisms that underpin this therapeutic pathway, are still unavailable. We hypothesize that 1) FMT from donors with limited presence of AR genes can be more effective than placebo in eradicating intestinal MDRB (focusing on carbapenem-resistant Enterobacteriaceae) and 2) microbial features of donors and patients can be reproducibly associated with clinical efficacy and clearance of AR genes. Our results will pave the way for the development of effective, targeted microbiome-based therapies against MDRB, alleviating the burden of AR, with considerable benefits for healthcare systems.

The extended aims of this study are:

* To identify FMT donors with limited presence of AR genes and store feces for FMT
* To assess the efficacy of FMT in eradicating intestinal MDRB (carbapenem-resistant Enterobacteriaceae) and collect stool samples for multi-omics analysis
* To characterize the fecal microbiome (bacteriome, virome, mycobiome), resistome, of donors and patients before and after FMT, to associate microbial profiles with clearance of AR genes and clinical efficacy, and identify the microbial features that influence it

The investigators will carry out a single-centre placebo-controlled, double blind randomised clinical trial of donor FMT vs placebo FMT in carriers of CRE Patients will be recruited among those referred to the infectious disease outpatient clinic of the Fondazione Policlinico Universitario "A. Gemelli". Patients with all inclusion criteria and none of the exclusion criteria (detailed in the specific section of this website) will be considered for this study.

Before randomisation, demographic data will be collected by the infectious disease staff. Moreover, patients will repeat rectal swab and stool culture.

Additionally, patients will be requested to give stool samples to be collected in a sterile, sealed container and stored at -80°C for metagenomic assessment of gut microbiome and meta-transcriptome assessment by the microbiology staff.

After baseline assessments, patients will be randomly assigned to one of the following treatment arms:

* Donor FMT (D-FMT)
* Placebo FMT (P-FMT) Patients in both groups will undergo a single FMT procedure by colonoscopy. Each patient in the donor FMT group will receive faeces from one single donor. Placebo FMT will be made of 250 mL water.

Donors will be recruited among healthy individuals, following international guidelines and according the new recommendation imposed by the reorganisation of faecal microbiota transplant during the COVID-19 pandemic. Only donors with a history of limited antibiotic usage (<5 antibiotic courses shorter than 10 days) will be chosen for resistome analysis, and only the three donors with the lowest rate of AR genes will be finally enrolled. Each donor will be asked to donate frequently (>7 aliquots/donor) and in a limited timeframe (3 months) to minimize the risk of changes in intestinal AR genes. Selected donors will be excluded if they will undergo antibiotic therapies within the donating period.

Thirty-six patients with intestinal colonization by CRE will be enrolled, based on sample size calculation. Informed consent will be collected from all patients. At baseline, stool samples will be collected for multi-omics analysis. Patients will be then randomized to colonoscopic FMT or placebo and will be followed up at week 1, 4 and 12 after treatments. At each visit they will undergo a clinical visit and a rectal swab for CRE, and stool samples will be collected and stored for multi-omics analysis.

Study Outcomes are detailed in the specific section of this website.

Statistical analysis will be performed both on an intention-to-treat and per-protocol basis. Differences among groups will be assessed with a two-tailed Wilcoxon-rank sum test for continuous data and with Fisher¿s exact probability test (using two- tailed P-values) for categorical data.

For microbiome analysis, statistical differences between group means will be calculated using a two-tailed Wilcoxon-Rank Sum Test, through the R statistical software package (R Core Team, Vienna, Austria).

Machine learning models will be used to identify and reproducibly characterize responder and nonresponder profiles. In particular, in a Python 3.9 environment using scikit-learn (ver. 0.22.1), two unsupervised ML algorithm, namely K-means and Agglomerative Hierarchical Clustering, will be used for creating patient clusters based on baseline microbiome features, in order to assess whether ML may identify distinct microbiome profiles associated with clinical response and changes in AR levels.

ELIGIBILITY:
Inclusion Criteria:

* >18 years;
* CRE diagnosed with rectal swab <15 days before evaluation;
* Ability to undergo study procedures and to give informed consent.

Exclusion Criteria:

* Active chronic gastrointestinal disorders;
* Previous colorectal surgery;
* Major comorbidities;
* Pregnancy/breastfeeding;
* Psychiatric disorders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
CRE eradication at week 4 after the end of treatments | 4 weeks
  The investigators will evaluate the number of participants who will obtain eradication of CRE carriage after treatments, at 4 weeks-follow-up, evaluated through rectal swab for CRE

SECONDARY OUTCOMES:
CRE eradication at week 1 and 12 after the end of treatments | 12 weeks
  The investigators will evaluate the number of participants who will obtain eradication of CRE carriage after treatments, at 1,2 and 12 weeks-follow-up, evaluated through rectal swab for CRE
microbiome changes after treatments | 12 weeks
  The investigators will evaluate microbiome changes through a multi-omic analysis (bacteriome, virome, mycobiome and resistome) . Biocomputational tools and unsupervised machine learning algorithms will be applied to identify microbial features (species, strains, genes, pathways, community structures) that are associated with longitudinal changes in gut resistome and clearance or persistence of AR genes, and link these dynamics to clinical response (eradication of CRE).

CONTACTS AND LOCATIONS:
Locations (1):
- Giovanni Cammarota, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers
Supporting Information: Study Protocol
Time Frame: data will be available after the completion of the study, for 5 years
Access Criteria: Data will be given upon reasonable request to the PI